CLINICAL TRIAL: NCT00064584
Title: Tolerability and PK/PD of Multiple Oral Doses of CT53518 in Patients With Acute Myelogenous Leukemia
Brief Title: Safety and Tolerance Study of Oral Doses of CT53518 to Treat Patients With Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-301
Record Dates: First submitted 2003-07-09; First posted 2003-07-10 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — tandutinib

INTERVENTIONS:
Drug: CT53518

SUMMARY:
This is the first study of the drug CT53518 when given to humans. The purpose of this study is to determine the highest dose of CT53518 that can safely be given to patients with Acute Myelogenous Leukemia (AML) and to identify the side effects associated with taking the drug. The study will evaluate how CT53518 is absorbed, broken down, and eliminated by the body. Additionally, the study will evaluate the effects of the drug on a specific type of cell in bone marrow and blood, known as a blast.

DETAILED DESCRIPTION:
This is a Phase 1, open label, dose escalating study at five clinical sites to determine dose limiting toxicity (DLT), maximum tolerated dose (MTD), pharmacokinetics, and the effect on the peripheral and bone marrow blast count of an oral 28-day course of CT53518 in patients with Acute Myelogenous Leukemia (AML) and myelodysplastic syndrome. This study will confirm the tolerability and assess the effects on the peripheral and bone marrow blast count of an oral 28-day course of CT53518 at or near the maximum tolerated dose in patients with AML displaying a specified mutation of the FLT-3 gene, internal tandem duplication (ITD).

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following inclusion criteria to be eligible to participate in the study.

* Men and women who are over 18 years of age and have one of the following conditions:

  * AML with relapse within 12 months of the completion of consolidation therapy who are not to receive gemtuzumab-ozogamicin; or
  * AML with relapse after 12 months of the completion of consolidation therapy for whom, in the opinion of the investigator, the risk of alternative therapy outweighs the possible benefit; or
  * newly diagnosed AML refractory to conventional remission-induction chemotherapy ("refractory" is defined as >10% blasts in blood and/or bone marrow upon recovery from two cycles of standard cytarabine-based induction chemotherapy); or
  * newly diagnosed, or previously treated AML, greater than 60 years of age and not or no longer a candidate for conventional remission-induction chemotherapy or gemtuzumab-ozogamicin
* No reproductive potential (surgically, post- menopausal, or using two methods of contraception)
* Demonstrated FLT-3 gene, internal tandem duplication mutation
* ECOG performance status of 0 to 2
* Has not received cytoreductive drug therapy for at least 4 weeks, and has not received hydroxyurea within 24 hours prior to first dose of the study drug
* Has not received a bone marrow transplant or peripheral blood stem cell transplant within the last two months
* Able to read and give written informed consent and has signed a consent form approved by the Investigator's Institutional Review Board (IRB)

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible to participate in the study:

* Participated in an investigational drug study in the last 30 days
* Serum Creatinine >2 mg/dL
* Evidence of a clinically significant liver disease by history, physical examination and/or laboratory data (e.g. transaminases exceeding 3 x ULN and/or total bilirubin > 2 mg/dL
* Known to have used illicit drugs within the last 30 days
* Has an uncontrolled active infection
* Pregnant or nursing mother
* Candidate for conventional chemotherapy (except hydroxyurea), including growth factors or hormonal therapy for cancer
* Any concomitant disease or condition which could interfere with or for which the treatment might interfere with the conduct of the study the, or which would, in the opinion of the Investigator and/or Sponsor, increase the risk of the patient's participation in the study. This includes but is not limited to alcoholism, drug dependency or abuse, psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-05; Primary Completion 2005-01 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon